CLINICAL TRIAL: NCT06493539
Title: A Novel Application of Closed Incision Negative Pressure Wound Therapy for the Post-Surgical Management of Lower Extremity Amputations: A Randomized Clinical Pilot Study
Brief Title: CiNPWT Lower Extremity Amputations (Closed Incision Neagtive Pressure Wound Therapy)
Acronym: CiNPWT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients recruited.
Sponsor: University of Southern California (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, David Armstrong, Dr. David Armstrong DPM, MD, PhD, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP-22-00260 USC
Record Dates: First submitted 2023-05-05; First posted 2024-07-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Wound Heal; Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Intervention
  Following amputation, at POD 1, CiNPWT will be applied in an "envelope-like" fashion, incorporating the incison line as well as ~10 cm of intact proximal residual limb tissue. The underlying skin will be protected with a contact layer and the negative pressure foam is applied for maximal surface area coverage. Negative pressure parameters are set to dynamic pressure control therapy (DPC) from -25 mmHg to -125 mmHg with a 2 minute on/2 minute off cycle and the dressing is left in place for three to five days.
  A patient may always be removed from treatment intervention whenever they wish.
  Control
  Following amputation, at POD 1, application of standard care (short stretch compression bandages and standard post-operative wound care) daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: Standard of Care (Active Comparator): Following amputation, at POD 1, application of standard care (short stretch compression bandages and standard post-operative wound care) daily.
  Interventions: Procedure: Standard of Care group
- CiNPWT treatment group (Experimental): Following amputation, at POD 1, CiNPWT will be applied in an "envelope-like" fashion, incorporating the incison line as well as ~10 cm of intact proximal residual limb tissue. The underlying skin will be protected with a contact layer and the negative pressure foam is applied for maximal surface area coverage. Negative pressure parameters are set to dynamic pressure control therapy (DPC) from -25 mmHg to -125 mmHg with a 2 minute on/2 minute off cycle and the dressing is left in place for three to five days.
  A patient may always be removed from treatment intervention whenever they wish.
  Interventions: Device: CINPWT

INTERVENTIONS:
Procedure: Standard of Care group — The control group will receive standard of care wound treatment
  Arms: Control group: Standard of Care
Device: CINPWT — Subject will receive CINPWT until discharged
  Arms: CiNPWT treatment group

SUMMARY:
The objective of this study is to evaluate prospectively the effect of a novel application of Closed Incision Negative Pressure Wound Therapy(CiNPWT), as delivered by the V.A.C. Ulta™ Therapy System (3M, USA) in individuals who have undergone a Lower Extremity Amputation(LEA) compared with standard of care compression wrapping and wound care post-LEA.

This a pilot-controlled exploratory trial including approximately 6-10 individuals who have undergone LEA (trans-metatarsal or higher) randomized between intervention (novel application of CiNPWT) and a control group (standard care).

DETAILED DESCRIPTION:
The objective of this study is to evaluate prospectively the effect of a novel application of Closed Incision Negative Pressure Wound Therapy (CiNPWT), as delivered by the V.A.C. Ulta™ Therapy System (3M, USA) in individuals who have undergone a Lower Extremity Amputation (LEA) compared with standard of care compression wrapping and wound care post-LEA.

Specific objectives:

1. Collect demographics and relevant data (e.g., risk factors and comorbidities) to compare intervention and control groups.
2. Measure post-surgical outcomes and compare both groups.

STUDY DESIGN

This a pilot-controlled exploratory trial including approximately 6-10 individuals who have undergone LEA (trans-metatarsal or higher) randomized between intervention (novel application of CiNPWT) and a control group (standard care).

DEVICE INFORMATION

The V.A.C. Ulta™ Therapy System (3M, USA) is a non-invasive wound closure system that uses controlled, localized negative pressure to promote healing in chronic and acute wounds. The subatmospheric (ie. negative) pressure system uses latex-free and sterile polyurethane or polyvinyl alcohol foam dressings that are individualized at the bedside to the appropriate size for every patient, and then covered with an adhesive drape to create an airtight seal. A SensaT.R.A.C.™ Pad directly contacts the foam dressing, and accurately senses, monitors, and maintains the target pressure at the wound site to provide controlled negative pressure. Tubing attached to the SensaT.R.A.C.™ Pad connects to a fluid collection canister contained in a programmable, portable, computer-controlled vacuum pump creating negative pressure at the wound surface interface.

Amputation (and revision/re-amputation) is a resection of a segment of a limb through a bone or through a joint.

Major amputation: Any resection proximal to the ankle.

Major amputation levels:

TT = transtibial amputation: amputation through the tibia and fibula (frequently referred to as "below knee amputation").

KD = knee disarticulation: amputation through the knee (frequently referred to as "through knee amputation").

TF = transfemoral amputation: amputation through the femur (frequently referred to as "above knee amputation").

Minor amputation: Any resection distal to the ankle.

Minor amputation levels:

TMA= transmetartarsal amputation.

The level will be determined using the electronic medical record of the patients and by the health care providers observations.

Wound dehiscence (partial or total) is a surgery complication where the incision reopens. Clinically reported by the health care providers. This will be also evaluated with digital photographs.

Infection at the surgical site and/or cellulitis of the residual limb are pathological states caused by invasion and multiplication of microorganisms in host tissues accompanied by tissue destruction and/or a host inflammatory response. This is usually based on soft tissue infection clinical criteria from Infectious Disease Society of America (IDSA) and will be reported by the health care provider.

Closed wound, defined as complete epithelialization at the surgical site, will be based on the health provider's clinical decision combined with medical record documentation. Determination is based on data from wound assessments and photographs performed by the treating clinician and documented in the Tissue Analytics wound imaging software. Photographs will be taken during patient visits (no more than 3x/wk) and if present, wound size, and tissue color percentages will be calculated by Tissue Analytics software. Any wound depth present will be measured manually by the treating therapist and entered into the Tissue Analytics system. Additional wound assessment characteristics that will be documented include periwound color and condition, drainage type or amount, and tissue type assessment. Agreement between clinician's documentation of closure and photographic measurements will be used to ascertain time to closure.

The tolerability/acceptability of CiNPWT will be measured:

* Pain which is a physical suffering or discomfort caused by CiNPWT is usually reported by the patient using the visual analogue scale at each visit.
* Anxiety about the treatment using Hamilton Anxiety Rating Scale (HAM-A)
* Quality of life using the Short Form-36 Questionaire

Baseline characteristics, risk factors and comorbidities will be extracted from the electronic medical record and validated with physical examination. Investigations can be done as necessary to complete missing data such as presence/absence of neuropathy, vascular status, etc., using best practice at the initial evaluation. As an example, blood samples will be obtained at the first evaluation to assess Hemoglobin A1c. If a patient is deemed at nutrition risk based on a nutrition screen done by nursing (Malnutrition Screening Tool), a dietitian will be consulted, and dietary supplementation will be initiated as needed.

All unscheduled or emergency visits will be listed.

At each encounter, the time to complete the treatment including dressings and compression (intervention and control) will be recorded by the clinician in the Electronic Medical Record.

ELIGIBILITY:
Inclusion criteria to select the participants (intervention and control):

* Individual aged 18 years or older
* Individual with a closed incision following LEA (transmetatarsal or proximal)
* Individual presents with adequate perfusion based on WIfI ischemia component score of less than 2 (>30mm Hg TCPO2 or higher at region of amputation)
* Individual presents with no residual surgical site infection (WIfI grade 0) post LEA
* Individual is competent to make their own medical decisions

Exclusion criteria (intervention and control):

* Individual presents with any defined contraindications to NPWT (e.g., allergy).
* Individual presents with residual acute osteomyelitis (after amputation).
* Individual with collagen vascular disease or malignant disease in the wound
* Individual has uncontrolled hyperglycemia (glycosylated hemoglobin [HbA1c]>12%).
* Individual is currently taking corticosteroids, immunosuppressive drugs, or chemotherapy and is not on stable course of therapy as determined by principal investigator
* Individual has a history of local radiation therapy that could impact the edema of the amputated limb.
* Individual has pre-existing conditions contributing to residual limb edema (i.e., nephropathy, congestive heart failure, primary lymphedema, etc.).

Withdrawal of individuals:

* Voluntary withdrawal
* Death
* Lost to follow-up
* Termination of compression therapy (control or intervention group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduction of edema as assessed using Girth measurements and Grading system. | Up to 8 weeks
  Measurement of edema reduction using the +1 to +4 grading system as well as girth measurements of lower extremity of using measuring tape.
Number of participants with Greater acceptability, tolerability and convenience as assessed by Short Form 36 and patient provided feedback. | Up to 8 weeks
  Determine the overall tolerability, acceptability, and convenience of the intervention using Patient surveys and patient provided feedback.
Number of participants with shorter time to ambulation and weight-bearing as measured by a stopwatch. | Up to 8 weeks
  CiNPWT effect on ambulation by measuring time to ambulation, time to weight-bearing as measured by a stopwatch.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0". | Up to 8 weeks
  CiNPWT on number of needed physical therapy visits, adverse events, surgical site infection, re-amputation/revision rate, dehiscence, dressing failure, unscheduled/emergency encounters, hospital-acquired pressure injuries.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fortington LV, Geertzen JH, van Netten JJ, Postema K, Rommers GM, Dijkstra PU. Short and long term mortality rates after a lower limb amputation. Eur J Vasc Endovasc Surg. 2013 Jul;46(1):124-31. doi: 10.1016/j.ejvs.2013.03.024. Epub 2013 Apr 28. PMID 23628328
- [Background] Low EE, Inkellis E, Morshed S. Complications and revision amputation following trauma-related lower limb loss. Injury. 2017 Feb;48(2):364-370. doi: 10.1016/j.injury.2016.11.019. Epub 2016 Nov 18. PMID 27890336
- [Background] Morisaki K, Yamaoka T, Iwasa K. Risk factors for wound complications and 30-day mortality after major lower limb amputations in patients with peripheral arterial disease. Vascular. 2018 Feb;26(1):12-17. doi: 10.1177/1708538117714197. Epub 2017 Jun 6. PMID 28587576
- [Background] Goldberg T. Postoperative management of lower extremity amputations. Phys Med Rehabil Clin N Am. 2006 Feb;17(1):173-80, vii. doi: 10.1016/j.pmr.2005.10.009. PMID 16517350
- [Background] Ahuja V, Thapa D, Ghai B. Strategies for prevention of lower limb post-amputation pain: A clinical narrative review. J Anaesthesiol Clin Pharmacol. 2018 Oct-Dec;34(4):439-449. doi: 10.4103/joacp.JOACP_126_17. PMID 30774224
- [Background] Nawijn SE, van der Linde H, Emmelot CH, Hofstad CJ. Stump management after trans-tibial amputation: a systematic review. Prosthet Orthot Int. 2005 Apr;29(1):13-26. doi: 10.1080/17461550500066832. PMID 16180374
- [Background] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Background] Scalise A, Calamita R, Tartaglione C, Pierangeli M, Bolletta E, Gioacchini M, Gesuita R, Di Benedetto G. Improving wound healing and preventing surgical site complications of closed surgical incisions: a possible role of Incisional Negative Pressure Wound Therapy. A systematic review of the literature. Int Wound J. 2016 Dec;13(6):1260-1281. doi: 10.1111/iwj.12492. Epub 2015 Oct 1. PMID 26424609
- [Background] Strugala V, Martin R. Meta-Analysis of Comparative Trials Evaluating a Prophylactic Single-Use Negative Pressure Wound Therapy System for the Prevention of Surgical Site Complications. Surg Infect (Larchmt). 2017 Oct;18(7):810-819. doi: 10.1089/sur.2017.156. Epub 2017 Sep 8. PMID 28885895
- [Background] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Background] Sanders JE, Fatone S. Residual limb volume change: systematic review of measurement and management. J Rehabil Res Dev. 2011;48(8):949-86. doi: 10.1682/jrrd.2010.09.0189. PMID 22068373
- [Background] Zwanenburg PR, Timmermans FW, Timmer AS, Middelkoop E, Tol BT, Lapid O, Obdeijn MC, Gans SL, Boermeester MA. A systematic review evaluating the influence of incisional Negative Pressure Wound Therapy on scarring. Wound Repair Regen. 2021 Jan;29(1):8-19. doi: 10.1111/wrr.12858. Epub 2020 Aug 21. PMID 32789902
- [Background] West J, Wetherhold J, Schulz S, Valerio I. A Novel Use of Next-Generation Closed Incision Negative Pressure Wound Therapy After Major Limb Amputation and Amputation Revision. Cureus. 2020 Sep 11;12(9):e10393. doi: 10.7759/cureus.10393. PMID 33062513
- [Background] Kilpadi DV, Olivie M. Evaluation of closed incision negative pressure therapy systems on the closure of incisional space model. J Wound Care. 2019 Dec 2;28(12):850-860. doi: 10.12968/jowc.2019.28.12.850. PMID 31825775
- [Background] Singh D, Livingstone JP, Lautze J, Murray PC. Measuring In-Vivo Foot Perfusion Distal to a Near-Circumferential Negative Pressure Wound Therapy Dressing via Thermal Imaging. Cureus. 2021 Sep 4;13(9):e17720. doi: 10.7759/cureus.17720. eCollection 2021 Sep. PMID 34650894
- [Background] Rafter N, Hickey A, Condell S, Conroy R, O'Connor P, Vaughan D, Williams D. Adverse events in healthcare: learning from mistakes. QJM. 2015 Apr;108(4):273-7. doi: 10.1093/qjmed/hcu145. Epub 2014 Jul 29. PMID 25078411
- [Background] van Netten JJ, Bus SA, Apelqvist J, Lipsky BA, Hinchliffe RJ, Game F, Rayman G, Lazzarini PA, Forsythe RO, Peters EJG, Senneville E, Vas P, Monteiro-Soares M, Schaper NC; International Working Group on the Diabetic Foot. Definitions and criteria for diabetic foot disease. Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3268. doi: 10.1002/dmrr.3268. Epub 2020 Jan 14. PMID 31943705
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E; Infectious Diseases Society of America. 2012 Infectious Diseases Society of America clinical practice guideline for the diagnosis and treatment of diabetic foot infections. Clin Infect Dis. 2012 Jun;54(12):e132-73. doi: 10.1093/cid/cis346. PMID 22619242
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Upton D, Stephens D, Andrews A. Patients' experiences of negative pressure wound therapy for the treatment of wounds: a review. J Wound Care. 2013 Jan;22(1):34-9. doi: 10.12968/jowc.2013.22.1.34. PMID 23299356
- [Background] Stouka X, Stergiannis P, Konstantinou E, Katsoulas T, Intas G, Skopa R, Fildissis G. Health-Related Quality of Life and Rehabilitation Costs of Patients with Amputated Limb. Adv Exp Med Biol. 2021;1337:237-243. doi: 10.1007/978-3-030-78771-4_27. PMID 34972911
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Result] Creager MA, Matsushita K, Arya S, Beckman JA, Duval S, Goodney PP, Gutierrez JAT, Kaufman JA, Joynt Maddox KE, Pollak AW, Pradhan AD, Whitsel LP. Reducing Nontraumatic Lower-Extremity Amputations by 20% by 2030: Time to Get to Our Feet: A Policy Statement From the American Heart Association. Circulation. 2021 Apr 27;143(17):e875-e891. doi: 10.1161/CIR.0000000000000967. Epub 2021 Mar 25. PMID 33761757
- [Result] Molina CS, Faulk J. Lower Extremity Amputation. 2022 Aug 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK546594/ PMID 31536201